CLINICAL TRIAL: NCT05959239
Title: Expanded Access With TB006 Treatment in Adults With Alzheimer's Disease and Related Dementias
Brief Title: TB006 Expanded Access (EA) Compassionate Use
Status: Available | Type: Expanded Access
Sponsor: TrueBinding, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TB006 EA Compassionate Use
Record Dates: First submitted 2023-07-14; First posted 2023-07-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Related Dementias; Expanded Access; TB006
MeSH Terms: conditions — Alzheimer Disease | interventions — TB006

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: TB006 — TB006 will be provided as single-use injectable glass vials.

SUMMARY:
This is an open-label, expanded access, compassionate use treatment protocol of TB006 treatment in participants who meet clinical diagnostic criteria for Alzheimer's disease (AD). Participants will receive TB006 at a dose of 4,000 milligrams (mg) intravenous (IV) over 1 hour every 28 days ± 5 days.

DETAILED DESCRIPTION:
A participant's physician who is interested in participating in this program will need to go to the company's website for further information and application forms.

ELIGIBILITY:
Inclusion criteria:

* Male and/or female participants > 55 years of age at the time of signing the informed consent.
* The participant is diagnosed with symptomatic AD or related dementia, meeting the clinical criteria for AD with an estimated or actual Mini-Mental State Examination (MMSE) score or 24 or less. All other medical conditions are stable and well managed. Clinical diagnosis of AD is consistent with the following:

  1. Probable AD, according to National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorder Association (NINCDS-ADRDA).
  2. Meets the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5) - Criteria for Major Neurocognitive Disorder (previously dementia).
* There must be clear documentation of the participant's declining cognitive and functional status, any and all treatments attempted, and response (or lack of) to treatments.
* The participant is not able to receive any of the current anti-AD medicines either due to intolerance or contraindication(s); or the participant's dementia has persistently declined despite receiving maximum allowable or tolerated doses of current anti-AD medicines, including aducanumab and lecanemab.
* The participant is unable or ineligible to enroll in another clinical trial for their condition. This is defined as:

  1. No ongoing trial for which the participant may qualify.
  2. An ongoing trial, but the participant does not qualify.
  3. No ongoing trial site within 50 miles of the participant's home.
* The investigator as well as the participant/caregiver must be informed of the potential risks and obligations of the program and decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the participant's medical history and program eligibility criteria. The participant, and/or, in the case of reduced decision-making capacity, the legally acceptable representative(s) consistent with national law and ethics approval is/are able to read, understand, and provide written informed consent.
* Has one (or more) identified adult program partner who either lives with the participant or has sufficient contact to provide assessment of changes in participant behavior and function over time and information on safety and tolerability; is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the clinic; agrees to accompany the participant to each program visit.
* Able to comply with the program procedures, including the ability to travel to the named clinic for monthly visits.

Exclusion criteria:

* Any clinically significant or uncontrolled medical condition, including but not limited to cardiovascular disease, respiratory disorder, malignancy, and hematology or clinical chemistry abnormality.
* Has undergone major surgery or experienced trauma in the last 14 days.
* Any condition or emergent intercurrent illness that, in the judgment of the investigator, could result in the risk of participation outweighing the potential benefit.
* Unable to comply with this program protocol or has health concerns that may increase risk, in the opinion of the investigator.
* Participated in a clinical trial with an investigation drug within the past 6 months.
* Enrolled in a previous TB006 clinical trial and either did not complete the clinical trial or had a significant treatment-related Adverse event (AE) that could cause an undue risk.

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Truebinding, Inc., Study Director — TrueBinding, Inc.

REFERENCES:
- See also: Related Info — https://truebinding.com/expanded-access